CLINICAL TRIAL: NCT00371423
Title: A Multi-center, Single-arm Study of the TAXUS Liberté™-SR Stent for the Direct Stenting Treatment of Patients With de Novo Coronary Artery Lesions
Brief Title: Direct Stenting of TAXUS Liberté™-SR Stent for the Treatment of Patients With de Novo Coronary Artery Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2032; TAXUS ATLAS Direct Stent
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Device: TAXUS Liberté™-SR
- Arm 2 (Other): Control data derived from ATLAS Workhorse Trial
  Interventions: Device: TAXUS Liberté™-SR

INTERVENTIONS:
Device: TAXUS Liberté™-SR — Paclitaxel-Eluting Coronary Stent System
  Arms: Arm 1
Device: TAXUS Liberté™-SR — Paclitaxel-Eluting Coronary Stent System
  Arms: Arm 2

SUMMARY:
TAXUS ATLAS Direct Stent is a global, multi-center, single-arm, noninferiority trial comparing results from patients in whom the TAXUS Liberté stent was directly implanted (direct stenting) versus results from patients in whom implantation with the TAXUS Liberté stent was preceded by balloon angioplasty (pre-dilatation). The Control group consists of patients in the main TAXUS ATLAS trial, in which pre-dilatation was mandatory. The primary objective is to compare outcomes of direct stenting with balloon catheter pre-dilatation. The primary hypothesis is that late outcomes with direct stenting of the TAXUS™ Liberté Paclitaxel-Eluting Coronary Stent System will be non-inferior to conventional implantation with balloon catheter pre-dilatation

ELIGIBILITY:
General Inclusion Criteria:

1. Patient is ≥18 years old.
2. Eligible for percutaneous coronary intervention (PCI)
3. Documented stable angina pectoris or unstable angina pectoris with documented ischemia, or documented silent ischemia
4. Left ventricular ejection fraction (LVEF) of ≥25%
5. Acceptable candidate for coronary artery bypass grafting (CABG)
6. Patient or legal guardian understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed
7. Willing to comply with all specified follow-up evaluations

Angiographic Inclusion Criteria:

1. Only one lesion appropriate for direct stenting (typically covered by one 24 mm stent or shorter), may be treated with the study stent. However, one additional lesion in a non-target vessel may be treated during the index procedure with a commercially available bare metal stent, heparin-coated stent or TAXUS Express stent.
2. Target lesion located within a single native coronary vessel
3. Target lesion enrolled for treatment may be composed of multiple lesions(not more than 10mm between diseased segments) but must be completely covered by one study stent.
4. Cumulative target lesion length is ≥10 mm and ≤28 mm (visual estimate) and is typically considered appropriate for direct stenting
5. RVD of ≥2.5 mm to ≤4.0 mm (visual estimate)
6. Target lesion diameter stenosis ≥50% (visual estimate)
7. Target lesion is de novo (i.e., a coronary lesion not previously treated)

General Exclusion Criteria:

1. Known hypersensitivity to paclitaxel
2. Any previous, concurrent or planned treatment with a non-study anti-restenotic drug-coated or drug-eluting coronary stent.
3. Previous or planned use of both the study stent and a non-study stent (i.e., commercial stent) in the treatment of the target vessel
4. Previous or planned treatment with intravascular brachytherapy in the target vessel
5. Planned CABG ≤9-months post-index procedure
6. MI within 72 hours prior to the index procedure and/or creatine kinase(CK) >2x the local laboratory's ULN unless CK-MB is <2x ULN.
7. Cerebrovascular Accident (CVA) within the past 6 months
8. Cardiogenic Shock
9. Acute or chronic renal dysfunction
10. Contraindication to ASA, or to both clopidogrel and ticlopidine
11. Patient is currently on warfarin or it is anticipated that treatment with warfarin will be required during any period within 6 months after the index procedure.
12. Leukopenia
13. Thrombocytopenia
14. Active peptic ulcer or active gastrointestinal (GI) bleeding
15. Known allergy to stainless steel
16. Any prior true anaphylactic reaction to contrast agents
17. Patient is currently, or has been treated with paclitaxel or other chemotherapeutic agents within 12-months of the index procedure
18. Anticipated treatment with paclitaxel or oral rapamycin during any period in the 9-months after the index procedure
19. Male or female with known intention to procreate within 3 months after the index procedure
20. Female of childbearing potential with a positive pregnancy test within 7 days before the index procedure, or lactating
21. Life expectancy of less than 24-months due to other medical condition
22. Co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
23. Currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.

Angiographic Exclusion Criteria:

1. Unprotected left main coronary artery disease (patient with protected left main disease can be enrolled only if the target lesion is in the RCA)
2. Target lesion is ostial in location (within 3.0 mm of vessel origin)
3. Target lesion and/or target vessel proximal to the target lesion is moderately or severely calcified by visual estimate
4. Target lesion and/or target vessel proximal to the target lesion is tortuous
5. Target lesion is located within or distal to a >60 degree bend in the vessel
6. Target lesion involves a bifurcation with a diseased (>50% stenotic)branch vessel >2.0 mm in diameter
7. Target lesion is totally occluded (TIMI flow<1) at baseline
8. Angiographic presence of probable or definite thrombus
9. Pre-treatment of the target vessel at the index procedure is not allowed with any device
10. A previously treated lesion within the target vessel:

    * <15 mm from the target lesion (visual estimate)
    * Performed </= 6 months from index procedure
    * >30% residual stenosis after previous treatment
11. Predilation with a balloon catheter of the target lesion and/or target vessel is not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2005-03; Primary Completion 2006-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Analysis segment percent diameter stenosis at 9-months | 9 Months

SECONDARY OUTCOMES:
Secondary Endpoints: Clinical procedural and technical success | 5 years
Utilization parameters (equipment utilization, procedure time, fluoroscopic time and amount of contrast used) | 9 Months
MACE rates at discharge, 1, 4 and 9-months and 1, 2, 3, 4, and 5 years post-index procedure | 5 Years
Stent thrombosis rate | 5 Years
Target Vessel Failure (TVF) | 5 Years
Target Vessel Revascularization (TVR) | 5 Years
QCA parameters (binary restenosis rate, in-stent %DS, MLD and late loss) | 9 Months
IVUS parameters (percent net volume obstruction, incomplete apposition, stent and area volumes, neointimal area volume) | 9 Months

CONTACTS AND LOCATIONS:
Overall Officials: John A Ormiston, MD, Principal Investigator — Mercy Hospital; Mark A Turco, MD, Principal Investigator — Washington Adventist Hospital; Peter Maurer, MPH, Study Director — Boston Scientific Corporation
Locations (25):
- United States (18):
  - University of Arkansas for Medical Sciences/Central Arkansas Veterans Healthcare Systems, Little Rock, Arkansas
  - Mercy General Hospital, Sacramento, California
  - University of California San Diego Medical Center, San Diego, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Florida Hospital, Orlando, Florida
  - St. Anthony's Medical Center, Rockford, Illinois
  - St. John's Hospital, Springfield, Illinois
  - The Heart Center, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Mary's Duluth Clinic Regional Heart Center, Duluth, Minnesota
  - Wake Medical Center, Raleigh, North Carolina
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - The Pennsylvania State University Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Northwest Cardiovascular Research Institute, Spokane, Washington
- New Zealand (4):
  - Mercy Angiography Unit, 98 Mountain Road, First Floor, Auckland, Epsom
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
- Singapore (2):
  - National University Hospital, Singapore
  - National Heart Centre, Singapore
- Shin Kong Memorial Hospital, Shih Lin Taipei, Taiwan

REFERENCES:
- [Derived] Ormiston JA, Charles O, Mann T, Hall JJ, McGarry T, Cannon LA, Webster MW, Mishkel GJ, Underwood PL, Dawkins KD. Final 5-year results of the TAXUS ATLAS, TAXUS ATLAS Small Vessel, and TAXUS ATLAS Long Lesion clinical trials of the TAXUS Liberte paclitaxel-eluting stent in de-novo coronary artery lesions. Coron Artery Dis. 2013 Jan;24(1):61-8. doi: 10.1097/MCA.0b013e32835b3932. PMID 23232250
- [Derived] Doi H, Maehara A, Mintz GS, Yu A, Wang H, Mandinov L, Popma JJ, Ellis SG, Grube E, Dawkins KD, Weissman NJ, Turco MA, Ormiston JA, Stone GW. Impact of post-intervention minimal stent area on 9-month follow-up patency of paclitaxel-eluting stents: an integrated intravascular ultrasound analysis from the TAXUS IV, V, and VI and TAXUS ATLAS Workhorse, Long Lesion, and Direct Stent Trials. JACC Cardiovasc Interv. 2009 Dec;2(12):1269-75. doi: 10.1016/j.jcin.2009.10.005. PMID 20129555
- [Derived] Mahmud E, Ormiston JA, Turco MA, Popma JJ, Weissman NJ, O'Shaughnessy CD, Mann T, Hall JJ, McGarry TF, Cannon LA, Webster MW, Mandinov L, Baim DS. TAXUS Liberte attenuates the risk of restenosis in patients with medically treated diabetes mellitus: results from the TAXUS ATLAS program. JACC Cardiovasc Interv. 2009 Mar;2(3):240-52. doi: 10.1016/j.jcin.2008.12.009. PMID 19463432
- [Derived] Ormiston JA, Mahmud E, Turco MA, Popma JJ, Weissman N, Cannon LA, Mann T, Lucca MJ, Lim ST, Hall JJ, McClean D, Dobies D, Mandinov L, Baim DS. Direct stenting with the TAXUS Liberte drug-eluting stent: results from the Taxus Atlas Direct Stent Study. JACC Cardiovasc Interv. 2008 Apr;1(2):150-60. doi: 10.1016/j.jcin.2008.01.003. PMID 19463293